CLINICAL TRIAL: NCT01743105
Title: Reproductibility of Time-motion-mode Ultrasound Diaphragm Measures in Patients With Acute Respiratory Distress in the Emergency Room
Brief Title: Reproductibility of TM-mode Ultrasound Diaphragm Measures in Patients With Acute Respiratory Distress in the ER
Acronym: EDDRA-Repro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2012/XBAC-01; 2012-A01094-39 (Other: RCB number); Bobbia EDDRA Repro (Other: BESPIM, Nîmes University Hospital)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: diaphragm movement; ultrasound; emergency room
MeSH Terms: conditions — Respiratory Distress Syndrome; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study population (Experimental): The study population consists of patients treated for acute respiratory distress in the emergency department at the Nîmes University Hospital. See inclusion and exclusion criteria.
  Interventions: Diaphragm excursion measures 1, Diaphragm excursion measures 2
  Interventions: Procedure: Diaphragm excursion measures 1; Procedure: Diaphragm excursion measures 2

INTERVENTIONS:
Procedure: Diaphragm excursion measures 1 — A first diaphragm ultrasound study will be carried out by investigator 1. A Vivid S6 GE Ultrasound will be used, with a phased array cardiac probe.
Procedure: Diaphragm excursion measures 2 — A second diaphragm ultrasound study will be carried out immediately after Ultrasound 1, and by investigator 2. The results are blinded between investigators. A Vivid S6 GE Ultrasound will be used, with a phased array cardiac probe.

SUMMARY:
The main objective of this study is to evaluate the inter-rater reproducibility of diaphragmatic excursion measures via time-motion-mode ultrasound (evaluation performed on the first measure) in patients experiencing acute respiratory distress emergencies.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* To assess the feasibility of measuring the diaphragmatic excursion in the context of emergency management (ratio of measured patients / included patients).
* To evaluate the time required for the measurement.
* To assess the intra-rater reproducibility of measurements of diaphragmatic excursion (comparison of first and second measures).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has acute respiratory distress defined by a respiratory rate > 25, and / or signs of struggle and hypoxia, oxygen saturation (SpO2) <90% and / or pH <7.35 and carbon dioxide partial pressure (pCO2) > 6 kPa (45 mm Hg)
* The patient breathes spontaneously (no respirator)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient or his/her representative refuses to sign the consent
* It is impossible to correctly inform the patient, or to correctly inform his/her representative
* The patient is pregnant, parturient, or breastfeeding
* The patient has a neurological or neuromuscular disease that modifies diaphragm function/movement; this does not include cases of decompensation (polyradiculoneuropathy, Lou Gehrig's disease, Myasthenia ...).
* Patient admitted with respiratory support treatment in progress
* Patient admitted with respiratory failure requiring immediate implementation of mechanical ventilation, thus preventing ultrasound measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01-27 (Actual); Study Completion 2014-01-27 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic excursion, first measure by investigator 1 | Baseline (day 0)
  in centimeters
Diaphragmatic excursion, first measure by investigator 2 | Baseline (day 0)
  in centimeters

SECONDARY OUTCOMES:
Time necessary to measure diaphragm movement amplitude (minutes) | Baseline (day 0)
Feasibility (yes/no) | Baseline (day 0)
  We were able to perform the required measurements (yes/no)
Diaphragmatic excursion, second measure by investigator 1 | Baseline (day 0)
  (centimeters)
Diaphragmatic excursion, second measure by investigator 2 | Baseline (day 0)
  (centimeters)

OTHER OUTCOMES:
Age | Baseline (day 0)
Sexe | Baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bobbia, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France

REFERENCES:
- [Result] Bobbia X, Clement A, Claret PG, Bastide S, Alonso S, Wagner P, Tison T, Muller L, de La Coussaye JE. Diaphragmatic excursion measurement in emergency patients with acute dyspnea: toward a new diagnostic tool? Am J Emerg Med. 2016 Aug;34(8):1653-7. doi: 10.1016/j.ajem.2016.05.055. Epub 2016 May 24. PMID 27251231